CLINICAL TRIAL: NCT02342041
Title: A Single-center, Double-blind, Placebo-controlled, Randomized, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SUVN-G3031 After Single Ascending Doses and Multiple Ascending Doses in Healthy Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of SUVN-G3031 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP13031H3
Record Dates: First submitted 2015-01-10; First posted 2015-01-19 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2015-09

CONDITIONS: Cognitive Disorders
Keywords: SUVN-G3031; histamine 3 (H3) receptor inverse agonist; first in human; safety; pharmacokinetics; tolerability; single dose; repeat dose
MeSH Terms: conditions — Cognitive Dysfunction | interventions — samelisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single ascending dose (Placebo Comparator): Single dose of SUVN-G3031or placebo in healthy male subjects
  Interventions: Drug: SUVN-G3031; Drug: Placebo
- Multiple ascending dose (Placebo Comparator): Multiple doses of SUVN-G3031 or placebo in healthy male subjects
  Interventions: Drug: SUVN-G3031; Drug: Placebo

INTERVENTIONS:
Drug: SUVN-G3031
Drug: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of SUVN-G3031 in healthy male subjects following single or multiple ascending doses.

DETAILED DESCRIPTION:
This is a single and multiple ascending dose study to assess the safety, tolerability and pharmacokinetics of SUVN-G3031 administered orally once a day to healthy male subjects. The study will be conducted under double-blind conditions.

The primary objective is to evaluate the safety and tolerability of SUVN-G3031 following oral administration of single or multiple ascending doses and estimate the maximum tolerated dose of SUVN-G3031, if possible.

The secondary objectives are to evaluate the single and repeat dose plasma pharmacokinetics following oral administration of single and multiple ascending doses of SUVN-G3031 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

• Healthy male aged 18 to 45 years with a BMI between 18 and 30 kg/m2, (inclusive).

Exclusion Criteria:

* Standard exclusion criterion for Phase 1 clinical trial in healthy subjects.
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs as judged by Investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single or multiple doses of SUVN-G3031 in healthy male subjects | Range of Day 1-19
  Safety variables - Adverse events, vital signs, electrocardiograms, telemetry, physical examination, and clinical laboratory assessments.

SECONDARY OUTCOMES:
Area under the SUVN-G3031 plasma concentration-time curve in a dosing interval (AUC0-tau) | Day 1
Area under the SUVN-G3031 plasma concentration-time curve from zero to infinity (AUC0-inf) | Day 14
Maximum observed concentration (Cmax) and time of observation (tmax) | Day 1 and Day 14
Oral clearance (CL/F), apparent volume of distribution (Vz/F), and elimination half life (t½) | Day 1 and Day 14
Accumulation index following multiple dosing of SUVN-G3031 (AI) | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Murtaugh Thomas, MD, Principal Investigator — Senior Medical Research Director
Locations (1):
- Quintiles, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Nirogi R, Mudigonda K, Bhyrapuneni G, Muddana NR, Shinde A, Goyal VK, Pandey SK, Mohammed AR, Ravula J, Jetta S, Palacharla VRC. Safety, Tolerability, and Pharmacokinetics of SUVN-G3031, a Novel Histamine-3 Receptor Inverse Agonist for the Treatment of Narcolepsy, in Healthy Human Subjects Following Single and Multiple Oral Doses. Clin Drug Investig. 2020 Jul;40(7):603-615. doi: 10.1007/s40261-020-00920-8. PMID 32399853